CLINICAL TRIAL: NCT02680210
Title: Self-defining Memories in Patients With a TBI and Their Relationships With Cognitive, Emotional and Behavioural Dimensions
Brief Title: Self-defining Memories in Patients With a TBI
Acronym: IDENTITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, AZOUVI, Principal investigator, Centre d'Investigation Clinique et Technologique 805
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A00996-43
Record Dates: First submitted 2016-01-29; First posted 2016-02-11 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Traumatic Brain Injuries; Neurobehavioral Manifestations; Cognition Disorders; Memory Deficits
MeSH Terms: conditions — Brain Injuries, Traumatic; Neurobehavioral Manifestations; Cognition Disorders; Memory Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cognitive measures and questionnaires (Other): the material of the study will consist of cognitive measures and questionnaires in order to (1) compare the cognitive performances and behavioral manifestations between patients with TBI and volunteers without neurological disorders and (2) to analyze the links between cognitive and behavioural measures in the TBI population
  Interventions: Other: Questionnaires and cognitive measures

INTERVENTIONS:
Other: Questionnaires and cognitive measures

SUMMARY:
The study will be conducted over 18 months. The main objective of this study is to explore the relationships between autobiographical memory and specific cognitive measures, as well as emotional and behavioural measures in patients who have suffered a moderate to severe TBI. Secondary objectives are to assess the psychometric properties of a self-defining memories questionnaire and to characterize autobiographical memory in the TBI population.

DETAILED DESCRIPTION:
A total of 40 participants (20 non-consecutive adults with a moderate or severe TBI and 20 volunteers with any history of neurological or psychiatric disease) will be recruited into the study. The duration of the protocol is 70 minutes. As regards the assessment, three questionnaires will be administered in order to evaluate self-defining memories, apathetic manifestations and anxio-depressive symptoms. In addition, four cognitive measures will be used to assess verbal episodic memory, working memory, cognitive flexibility and verbal fluency.

ELIGIBILITY:
Inclusion Criteria:

* patients with a moderate or severe TBI occurred at least 6 months ago (initial Glasgow Coma Scale score ≤ 12 or post-traumatic amnesia duration > 1 week)
* patients ≥ 18 years old and who have signed a letter of information

Exclusion Criteria:

* history of neurological and/or psychiatric disease
* persistent motor, sensitive and instrumental disorders that could disturb the efficient evaluation of the participant
* patients who refused to participate in the study
* non affiliation to a social security scheme
* patients under guardianship or trusteeship
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
self-defining memory score | 20 minutes
  self-defining memories will be measured using the self-defining memories questionnaire

SECONDARY OUTCOMES:
verbal episodic memory score | 20 minutes
  verbal episodic memory will be measured using the California Verbal Learning Test
working memory score | 10 minutes
  working memory will be measured using verbal span task
cognitive flexibility score | 5 minutes
  cognitive flexibility will be measured using the Trail Making Test
verbal fluency score | 5 minutes
  verbal fluency will be measured using the verbal fluency task
apathy score | 5 minutes
  apathetic manifestations will be measured using the Apathy Evaluation Scale
anxio-depressive score | 5 minutes
  anxio-depressive symptoms will be measured using the Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Annabelle Arnould, psychologue, Study Chair — Hôpital Raymond Poincaré
Locations (1):
- Hôpital Raymond Poincaré, Garches, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No